CLINICAL TRIAL: NCT03176745
Title: Determination of the Optimal Number of Multiple Breath Washout Tests in Adults With Pulmonary Disease and Healthy Controls
Brief Title: Number of Multiple Breath Washout Tests in Adults With Pulmonary Disease and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: MBW-number
Record Dates: First submitted 2017-06-02; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Healthy Controls; Chronic Obstructive Pulmonary Disease; Bronchial Asthma; Sarcoidosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy controls: * no history of pulmonary disease
  * absence of symptoms, smoking history < 10 pack years
  * normal lung function testing
  Interventions: Diagnostic Test: multiple breath washout
- chronic obstructive pulmonary disease: * clinical history and/or specialist diagnosis of COPD and risk factor(s)
  * persistent bronchial obstruction and/or hyperinflation and/or radiological sign of emphysema, each without alternative explanation
  * dyspnea, cough and/or sputum production
  Interventions: Diagnostic Test: multiple breath washout
- bronchial asthma: * clinical history and/or specialist diagnosis of bronchial asthma
  * respiratory symptoms compatible with asthma varying over time
  * variable and/or reversible obstructive ventilation disorder and/or airway hyperresponsiveness
  * exclusion of alternative explanation
  Interventions: Diagnostic Test: multiple breath washout
- sarcoidosis: * clinical history and/or specialist diagnosis of sarcoidosis
  * lymphocytic alveolitis and CD4/CD8 > 3.5 in bronchoalveolar lavage and/or noncaseating epithelioid granuloma
  * exclusion of alternative explanation
  Interventions: Diagnostic Test: multiple breath washout

INTERVENTIONS:
Diagnostic Test: multiple breath washout — determination of lung clearance index using SF6 multiple breath washout

SUMMARY:
The investigators aim to determine the optimal number of measurements required for multiple-breath-washout derived lung function parameters in adults with pulmonary disease as well as in healthy controls

ELIGIBILITY:
Inclusion criteria:

- informed consent

Exclusion Criteria:

* inability to perform multiple breath washout testing

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: inpatients, outpatients, students, employees
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
change of lung clearance index (LCI) as determined by multiple breath washout | 60 minutes
  comparing the repeatability of duplicate vs. triplicate LCI measurements

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trinkmann F, Gotzmann J, Saur D, Schroeter M, Roth K, Stach K, Borggrefe M, Saur J, Akin I, Michels JD. Multiple breath washout testing in adults with pulmonary disease and healthy controls - can fewer measurements eventually be more? BMC Pulm Med. 2017 Dec 11;17(1):185. doi: 10.1186/s12890-017-0543-y. PMID 29228942